CLINICAL TRIAL: NCT05414084
Title: Identification of Aggregate Metabolic Phenotypes for the Main Dietary (Poly)Phenols and Assessment of the Factors Associated With Their Formation: Development of an Oral (Poly)Phenol Challenge Test (OPCT)
Brief Title: Aggregate Metabolic Phenotypes for (Poly)Phenols: Development of an Oral (Poly)Phenol Challenge Test (OPCT)
Acronym: OPCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliero-Universitaria di Parma (Other); University of Birmingham (Other); National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Pedro M. Mena Parreño, Doctor, University of Parma
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1352/2020/SPER/UNIPR
Record Dates: First submitted 2022-05-26; First posted 2022-06-10 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2024-02

CONDITIONS: Individual Variability in (Poly)Phenol Metabolism; Cardiometabolic Health
Keywords: intervention study; (poly)phenols; metabolic phenotypes; metabotypes; cardiometabolic diseases; inter-individual variability; phenolic metabolites

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- (Poly)phenol tablets (Experimental): Single ingestion of 3 tablets containing different amounts of the most representative dietary (poly)phenols (i.e. flavonoid subclasses, phenolic acids, lignans, ellagitannins, stilbenes, flavonols, procyanidins and phenylethanoids)
  Interventions: Dietary Supplement: Oral (poly)phenol challenge test (OPCT)

INTERVENTIONS:
Dietary Supplement: Oral (poly)phenol challenge test (OPCT) — Nutritional challenge with standardized (poly)phenol-rich tablets

SUMMARY:
The study is a single-dose acute clinical trial aiming at identifying aggregate metabolic phenotypes for the main dietary (poly)phenols and assessing the factors associated with their formation.

The treatment consists of a nutritional challenge representative of the consumption of (poly)phenols in Europeans (so-called oral (poly)phenol challenge test, OPCT) and foresees the supplementation of three standardized tablets rich in (poly)phenols, prepared from various commercially available plant extracts constituting sources of specific (poly)phenols. Urinary excretion of (poly)phenol metabolites will be evaluated at 24 hours after tablet consumption or, for two subgroups of volunteers, at different time points for 24 hours upon tablet consumption. Blood pressure and heart rate will also be measured and anthropometric data collected. Information will be collected on genetic polymorphisms related to the metabolism of (poly)phenols, gene expression, standard cardiometabolic health biomarkers, cardiometabolic risk scores and gut microbiota profile, through the collection of urine, blood and stool samples. Volunteers will follow a (poly)phenol-free diet before and after the OPCT. To check compliance with food restrictions, a 24-hour recall will be carried out on each visit. For a sub-group of 50 subjects, 3 months after the first challenge, the OPCT will be repeated with further urinary and fecal collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-74 y)
* BMI 18.5-35 kg/m^2

Exclusion Criteria:

* Past cardiovascular events and metabolic diseases including diabetes
* Inflammatory bowel diseases or gastro-intestinal surgery
* Renal (GFR<60 ml/min) or hepatic diseases (liver enzymes >2.5 fold higher)
* Immunodeficiency or autoimmune diseases (other than well-compensated hypothyroidism)
* Mental disorders
* Antibiotic therapy within the last month
* Food allergies
* Pregnancy or lactation

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Identification of aggregate phenolic metabotypes | 24 hours post-consumption
  Assessing the variability in the urinary excretion of phenolic metabolites among volunteers after consumption of (poly)phenol-rich tablets by using data-driven clustering.

SECONDARY OUTCOMES:
Assessing common cardiometabolic health biomarkers in blood samples | Baseline
  Samples will be processed for the analysis of common biomarkers of cardiometabolic health: total cholesterol (mg/dL), HDL-cholesterol (mg/dL), triglycerides (mg/dL), glucose (mg/dL), insuline (uUI/mL). Analyses will follow standardised routine procedures.
Assessing risk prediction scores | Baseline
  Risk prediction scores (i.e., Framingham General Cardiovascular Risk Score, Framingham Heart Study Primary Risk Functions for heart disease, stroke, diabetes, fatty liver disease, and hypertension, Atherosclerotic Cardiovascular Disease (ASCVD) Risk, QRISK3®, QDScore®, Finnish Diabetes Risk Score (FINDRISC)) will be assessed to understand their relationship with the aggregate phenolic metabotypes observed. The higher the scores, the worse the risk of developing the disease.
Evaluating trimethylamine N-oxide (TMAO) in urine and plasma samples | Baseline
  TMAO will be quantified in baseline urine and fasting plasma samples by UHPLC-MS/MS.
Evaluating eicosanoids in urine samples | Baseline
  Eicosanoids, including prostaglandins, thromboxanes, leukotrienes, isoprostanes and neuroprostanes will be evaluated in baseline urine samples (0-h) by UHPLC-QqQ-MS/MS.
Assessing DNA oxidation catabolites and branched fatty acyl esters of hydroxyl fatty acids (FAHFAs) in plasma samples | Baseline
  DNA oxidation catabolites and FAHFAs will be measured in fasting plasma samples by UHPLC-QqQ-MS/MS.
Determining genetic differences among subjects | Baseline
  Genotyping will be conducted using genome wide, SNP array approach untargeted methodology, using commercially available SNP arrays and a tSNP approach. This approach will involve the genotyping of approximately 300 SNPs. Genomic DNA will be prepared from PBMCs isolated from blood samples.
Assessing transcriptomic signatures in peripheral blood mononuclear cells (PBMCs). | Baseline
  Specific patterns of gene expression related to each metabotype will be investigated in PBMCs by using a microarray-based approach. Analysis will be carried out in a subset of 10 samples for each metabotype.
Determining gut microbiota composition and functionality in fecal samples | Baseline
  Microbial profiling will be assessed by shallow shotgun metagenomics. Full shotgun metagenomics analysis will be carried out to determine functional pathways in a sample subset (50 samples).
Assessing dietary habits | Baseline
  Dietary habits will be assessed through a food frequency questionnaire.
Assessing anthropometric measurements | Baseline
  Weight and height will be combined to report BMI in kg/m^2 and this will be carried out according to standardized procedures. Waist circumference and hip circumference, waist-to-height ratio, waist-to-hip ratio, and body composition measurement (skinfold test and bioelectrical impedance analysis).
Assessing blood pressure and heart rate | Baseline
  Systolic and diastolic blood pressure and heart rate of each volunteer will be obtained after a 5-min rest in a seated position in the baseline visit.
Evolution over the time of the phenolic metabolites in urine samples | Different collection times for 24 hours (0; 0-3; 3-6; 6-9; 9-12; 12-24; 24 h)
  Assessed by using UHPLC-MS/MS for individual detection and quantification.
Untargeted urinary metabolomics | Baseline and 24 hours post-consumption
  The untargeted LC-IMS-MS metabolomics approach will allow to assess potential differences among the metabolomes of individuals belonging to different aggregate phenolic metabotypes.
Assessing the stability of aggregate phenolic metabotypes among individuals after 3 months | 24 hours post-consumption in a test carried out after 3 months after the first supplementation
  Assessing the variability in the urinary excretion of phenolic metabolites among volunteers after consumption of (poly)phenol-rich tablets, considering the metabotype to which each volunteer belongs to once the volunteer re-do the oral (poly)phenol challenge test after 3 months from the first supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro M Mena Parreño, PhD, Principal Investigator — University of Parma
Locations (2):
- Italy (2):
  - University of Parma - Plesso Biotecnologico Integrato, Parma, PR
  - Azienda Ospedaliero-Universitaria di Parma, Parma, PR

IPD SHARING:
Plan to Share IPD: No